CLINICAL TRIAL: NCT00518869
Title: Complementary Treatment of PG2 to Improve Clinical Benefit Response and Quality of Life in Fatigue
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP010
Record Dates: First submitted 2007-08-18; First posted 2007-08-21 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Quality of Life; Fatigue; Complementary
Keywords: Non-Small Cell Lung Cancer (NSCLC); Complementary and Alternative Medicine (CAM); Chemotherapy; Myelosuppression; Quality of Life; Fatigue; EORTC QLQ-C30 and LC13
MeSH Terms: conditions — Fatigue; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): PG2 plus standard chemotherapies
  Interventions: Drug: PG2
- Placeo group (Placebo Comparator): Placebo plus standard chemotherapies
  Interventions: Drug: PG2

INTERVENTIONS:
Drug: PG2 — 500 mg PG2 / 500 ml normal saline IV infusion for 3 hours once daily for 4 doses in the 1st week, 3 doses in the 2nd week and 3 doses in the 3rd week of each chemo-cycle for three cycles. Total 10 doses will be given in each cycle even with skip days.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of PG2 as a complementary treatment to conventional chemotherapy among NSCLC patients. In reference to previous studies, "Clinical Benefit Response" and "Incidence of Grade III plus VI Neutropenia" will be used as the primary endpoints in this study. Clinical Benefit Response is a metric measurement including change in cancer or cancer treatment related "fatigue" which is related to chronic fatigue syndrome (CFS), change in karnofsky performance status and change in weight. The secondary endpoints include patient's global quality of life, and the blood c-reactive protein level which is related to weight change, tumor response, survival time, incidences of myelosuppression (including neutropenia, anemia and thrombocytopenia) and the related G-CSF and antibiotics consumption.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized and placebo-controlled study to evaluate complementary effect of PG2 in patients with advanced non-small-cell lung cancer under conventional chemotherapy. Patients with Stage IIIb-IV non-small-cell lung cancer will be screened by inclusion and exclusion criteria and only eligible patients will be enrolled into this study.

All enrolled patients will be randomized to PG2 or Placebo arm and will receive the cisplatin-based chemotherapy treatment (Cisplatin 75mg/m2 and Docetaxel 60mg/m2 on Day1) during the first three 21-day chemo-cycles. Chemo regimen modification is allowable, as usual, in case of disease progression or unacceptable toxicity (see Section 6). After randomization, each patient will be administered with PG2 or placebo for 4 days in the 1st week, 3 days in the 2nd week and 3 days in the 3rd week of each chemo-cycle for 3 cycles (Dosing Schedule in Section 6). Total 10 doses will be given in each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form.
* 18 ~ 75 years old
* Locally advanced or metastatic with inoperable stage IIIb-IV non-small-cell lung cancer.
* Chemo/Radio naive patient
* Karnofsky Performance Scores ≧ 70.
* Adequate bone marrow reserve.
* Adequate liver function.
* Adequate renal function.
* Women with childbearing potential are willing to take contraception measures through the whole treatment course.
* Life expectancy ≧ 3 months
* Patient must be willing and able to complete quality of life questionnaires.

Exclusion Criteria:

* Female patients are pregnant or breast-feeding
* Patients have brain metastases, stroke or major psychiatric disease.
* Patients with uncontrolled systemic disease such as active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus.
* Patients have enrolled or have not yet completed other investigational drug trials within 30 days before randomization.

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Response | within and between each chemo-cycle (21 days)
Incidence of Grade III plus IV Neutropenia | within and between each chemo-cycle (21 days)

SECONDARY OUTCOMES:
Quality of Life Assessments | within and between each chemo-cycle (21 days)
The blood c-reactive protein level which is related to weight change | within and between each chemo-cycle (21 days)
Tumor Response | 3 months
Survival Time | one year
Incidences of myelosuppression and the related G-CSF consumption and antibiotics consumption | within and beween each chemo-cycle (21 days)

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Chang-Gung Memorial Hospital - Kaoshiung, Kaohsiung City
  - Kaoshiung Medical University Hospital, Kaohsiung City
  - Chang-Gung Memorial Hospital, Linkou, Linkou District
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei